CLINICAL TRIAL: NCT03158532
Title: Prevention of Radial Artery Occlusion After Transradial Access Using Nitroglycerin
Acronym: Patens
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto de Cardiologia de Santa Catarina (Other)
Responsible Party: Principal Investigator, Roberto Léo da Silva, Intervencional cardiologist, Instituto de Cardiologia de Santa Catarina
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Nitroglycerin on Occlusion
Record Dates: First submitted 2017-05-16; First posted 2017-05-18 (Actual); Results first posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Injury of Radial Artery
MeSH Terms: interventions — Nitroglycerin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo I/Placebo II (Placebo Comparator): 0,9% Saline 10 mL was given intra-arterially through the sheath at the start of a transradial procedure (right after sheath placement) and 0,9% Saline 10 mL was given intra-arterially through the sheath at the end of procedure (just before sheath removal).
  Interventions: Drug: Placebo I; Drug: Placebo II
- Nitroglycerin I/Placebo II (Experimental): 500 microgram of Nitroglycerin (in 10 mL saline) was given intra-arterially through the sheath at the start of a transradial procedure (right after sheath placement) and 0,9% Saline 10 mL was given intra-arterially through the sheath at the end of procedure (just before sheath removal).
  Interventions: Drug: Nitroglycerin I; Drug: Placebo II
- Placebo I /Nitroglycerin II (Active Comparator): 0,9% Saline 10 mL was given intra-arterially through the sheath at the start of a transradial procedure (right after sheath placement) and 500 microgram of Nitroglycerin (in 10 mL saline) was given intra-arterially through the sheath at the end of procedure (just before sheath removal).
  Interventions: Drug: Placebo I; Drug: Nitroglycerin II
- Nitroglycerin I /Nitroglycerin II (Experimental): 500 microgram of Nitroglycerin (in 10 mL saline) was given intra-arterially through the sheath at the start of a transradial procedure (right after sheath placement) and 500 microgram of Nitroglycerin (in 10 mL saline) was given intra-arterially through the sheath at the end of procedure (just before sheath removal).
  Interventions: Drug: Nitroglycerin I; Drug: Nitroglycerin II

INTERVENTIONS:
Drug: Nitroglycerin I — 500 microgram of Nitroglycerin intra-arterially administered through the radial sheath, right after sheath placement and before catheterization.
  Other Names: Tridil
  Arms: Nitroglycerin I /Nitroglycerin II; Nitroglycerin I/Placebo II
Drug: Placebo I — Saline 0,9% intra-arterially administered through the radial sheath, right after sheath placement and before catheterization.
  Other Names: Saline
  Arms: Placebo I /Nitroglycerin II; Placebo I/Placebo II
Drug: Nitroglycerin II — 500 microgram of Nitroglycerin intra-arterially administered through the radial sheath, just before sheath removal and before hemostasis.
  Other Names: Tridil
  Arms: Nitroglycerin I /Nitroglycerin II; Placebo I /Nitroglycerin II
Drug: Placebo II — Saline 0,9% intra-arterially administered through the radial sheath, just before sheath removal and before hemostasis.
  Other Names: Saline
  Arms: Nitroglycerin I/Placebo II; Placebo I/Placebo II

SUMMARY:
The radial approach for a coronary angiography has became popular in several centers because of its simplicity and fewer complications. The radial artery occlusion (RAO) is the main inconvenient and impose a limitation of future use of the radial artery as an access site for catheterization in the future. Several strategies have been used to decrease the incidence of RAO (heparin, patent hemostasis, etc). Nitrates in intra-arterial have been widely studied in prevention of this spasm. Current data show that nitroglycerin intra-arterial at the end of the procedure reduce the incidence of RAO. The hypothesis that use of nitroglycerin at the start of catheterization would have the same effect was not tested.

DETAILED DESCRIPTION:
Transradial access (TRA) has been increasingly adopted for diagnostic and interventional cardiovascular procedures in many centers worldwide. This is largely driven by the evidence supporting an unequivocal reduction in access site-related complications associated with TRA compared with transfemoral access, as well as reduction in cost and increased patient comfort. The radial artery occlusion (RAO) is the main inconvenient and impose a limitation of future use of the radial artery as an access site for catheterization in the future. RAO is the most commun complication of transradial access, and its incidence continues to reach up to 12%.

Nitrates in intra-arterial have been widely studied in prevention of this spasm. Nitroglycerin binds to the surface of endothelial cells and undergoes two chemical reductions to form nitric oxide (NO). The nitric oxide then moves out of the endothelial cell and into an adjacent smooth muscle cell, where it promotes the formation of cyclic guanosine monophosphate (cGMP), which then promotes muscle relaxation. Current data show that nitroglycerin intra-arterial at the end of the procedure reduce the incidence of radial artery occlusion.

A big sheath to artery size ratio could reduce the incidence of RAO, so the main objective of this study is to evaluate whether administration of nitroglycerin at the start of a transradial procedure may preserve the patency of the radial artery; as well, confirm if nitroglycerin administration just before sheet removal helps to keep the radial artery patency.

ELIGIBILITY:
Inclusion Criteria:

* Indication for cardiac catheterization;
* Suitable candidates for transradial approach;
* Use of 5 or 6 French sheath in the procedure;
* Signed informed consent.

Exclusion Criteria:

* Unable to tolerate nitrates or known allergy to nitrates;
* Use of any nitrate, by any route of administration, up to 1 hour before the procedure;
* ST-segment elevation acute myocardial infarction patients during the first 12 hours of sympton onset;
* Intubated patients (on mechanical ventilation);
* Complications before or during procedure (cardiac arrest, pulmonary edema, cardiogenic shock, stroke);
* Prior inclusion in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2040 (Actual)
Dates: Start 2017-07-06 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roberto L da Silva, MD, Study Chair — Instituto de Cardiologia de Santa Catarina; José R Costa Júnior, PhD, Study Director — Instituto Dante Pazzanese de Cardiologia
Locations (3):
- Brazil (3):
  - Hospital Universitário Professor Polydoro Ernani de São Thiago, Florianópolis, Santa Catarina
  - Instituto de Cardiologia de Santa Catarina, São Jose, Santa Catarina
  - Irmandade Santa Casa Misericórdia Marília, Marília, São Paulo

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo I/Placebo II | Nitroglycerin I/Placebo II | Placebo I /Nitroglycerin II | Nitroglycerin I /Nitroglycerin II
Started | 510 | 510 | 510 | 510
Completed | 510 | 510 | 510 | 510
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo I/Placebo II | Nitroglycerin I/Placebo II | Placebo I /Nitroglycerin II | Nitroglycerin I /Nitroglycerin II | Total
Number analyzed (Participants) | 510 | 510 | 510 | 510 | 2040
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.52 (10.35) | 62.06 (10.29) | 61.52 (10.35) | 62.06 (10.29) | 61.79 (10.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 188 | 199 | 199 | 188 | 774
  Male | 322 | 311 | 311 | 322 | 1266
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Radial Artery Occlusion
Description: Incidence of radial artery occlusion as confirmed by absence of antegrade flow in vascular doppler ultrasound
Time Frame: 2 to 24 hours after procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo I/Placebo II | Nitroglycerin I/Placebo II | Placebo I /Nitroglycerin II | Nitroglycerin I /Nitroglycerin II
Number analyzed (Participants) | 510 | 510 | 510 | 510
Participants | 13 | 13 | 10 | 13

2. Secondary Outcome: Late Radial Artery Occlusion
Description: Incidence of radial artery occlusion as confirmed by absence of antegrade flow in vascular doppler ultrasound
Time Frame: 30 days after procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo I/Placebo II | Nitroglycerin I/Placebo II | Placebo I /Nitroglycerin II | Nitroglycerin I /Nitroglycerin II
Number analyzed (Participants) | 510 | 510 | 510 | 510
Participants | 9 | 9 | 7 | 9

3. Secondary Outcome: Pain Assessment
Description: Pain felt by the patient in the forearm, assessed using numeric pain rating scale ranging from 0 to 10, 0 best (no pain) 10 worst (unbearable pain)
Time Frame: up to 24 hours after procedure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo I/Placebo II | Nitroglycerin I/Placebo II | Placebo I /Nitroglycerin II | Nitroglycerin I /Nitroglycerin II
Number analyzed (Participants) | 510 | 510 | 510 | 510
score on a scale | 2.7 (.42) | 2.4 (.37) | 2.7 (.42) | 2.4 (.37)

4. Secondary Outcome: Spasm (Operator Evaluation)
Description: Catheter friction, as experienced by the operator (subjective measure), during the realization of the procedure
Time Frame: During the realization of the procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo I/Placebo II | Nitroglycerin I/Placebo II | Placebo I /Nitroglycerin II | Nitroglycerin I /Nitroglycerin II
Number analyzed (Participants) | 510 | 510 | 510 | 510
Participants | 12 | 10 | 10 | 12

5. Secondary Outcome: Procedure Duration
Description: Total duration of the procedure in seconds, from puncture to haemostatic dressing.
Time Frame: Duration of the procedure
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Placebo I/Placebo II | Nitroglycerin I/Placebo II | Placebo I /Nitroglycerin II | Nitroglycerin I /Nitroglycerin II
Number analyzed (Participants) | 510 | 510 | 510 | 510
seconds | 1,193.22 (1,105.82) | 1,216.29 (1,179.52) | 1,229.83 (1,208.30) | 1,179.67 (1,073.80)

6. Secondary Outcome: Radiation Exposure
Description: Total radiation used in the procedure
Time Frame: During the procedure
Measure: Mean (Standard Deviation); unit: mGy
Arm/Group | Placebo I/Placebo II | Nitroglycerin I/Placebo II | Placebo I /Nitroglycerin II | Nitroglycerin I /Nitroglycerin II
Number analyzed (Participants) | 510 | 510 | 510 | 510
mGy | 584.52 (497.54) | 591.30 (524.38) | 599.78 (559.61) | 576.09 (457.49)

ADVERSE EVENTS:
Time Frame: 30 days
Description: Hand isquemia
Arm/Group | Placebo I/Placebo II | Nitroglycerin I/Placebo II | Placebo I /Nitroglycerin II | Nitroglycerin I /Nitroglycerin II
All-Cause Mortality (participants affected / at risk) | 0/510 | 0/510 | 0/510 | 0/510
Serious Adverse Events (participants affected / at risk) | 0/510 | 0/510 | 0/510 | 0/510
Other Adverse Events (participants affected / at risk) | 6/510 | 12/510 | 6/510 | 13/510
OTHER ADVERSE EVENTS (reported when occurring in more than 1.8% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo I/Placebo II (N=510) | Nitroglycerin I/Placebo II (N=510) | Placebo I /Nitroglycerin II (N=510) | Nitroglycerin I /Nitroglycerin II (N=510)
Hypotension (Cardiac disorders) | 6 (6) | 12 (12) | 6 (6) | 13 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-12-04): https://cdn.clinicaltrials.gov/large-docs/32/NCT03158532/Prot_SAP_000.pdf